CLINICAL TRIAL: NCT01889290
Title: Pharmacokinetics of Once Daily Subcutaneous Methylnaltrexone in Neurointensive Care Patients With High Dose Sufentanil Analgosedation
Brief Title: Methylnaltrexone Pharmacokinetics in Neurointensive Care Patients
Acronym: RELZH12
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELZH12
Record Dates: First submitted 2013-06-17; First posted 2013-06-28 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Opioid Use, Unspecified With Other Opioid-induced Disorder
Keywords: methylnaltrexone; opioid-antagonist; Obstipation; pharmacokinetics
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylnaltrexone (Experimental): Pharmacokinetics of methylnaltrexone administered once daily
  Interventions: Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Methylnaltrexone — Methylnaltrexone 12mg s.c. administered once daily until treatment stop of sufentanyl
  Other Names: Relistor

SUMMARY:
* Assessment of pharmacokinetic parameters of once daily subcutaneously administered methylnaltrexone in 10 evaluable neurointensive care patients.
* Quantification of methylnaltrexone passage through the blood-brain-barrier in critically ill patients with severe cerebral affections.
* Observation of laxation response after methylnaltrexone application and relation to plasma concentrations of methylnaltrexone.
* Assessing the safety of once daily administered methylnaltrexone in neurointensive care patients.
* Trial with medicinal product

DETAILED DESCRIPTION:
After administration of methylnaltrexone s.c. multiple peripheral blood samples and additionally two liquor samples are drawn during a dose interval on day 1, 3, and 5 of drug administration.

ELIGIBILITY:
Inclusion criteria:

* hospitalisation in the neurointensive care unit
* deep sedation with sufentanil doses of = 40 mcg/h
* male or female aged 18 years or older
* females: negative pregnancy test
* Ventricular drainage as part of needed therapeutic measures

Exclusion criteria:

* History of hypersensitivity to methylnaltrexone (Relistor®)
* confirmed or suspected obstructive ileus or factors possibly leading to intestinal obstruction (e.g. an intestinal tumor)
* increased risk for patients with localized or diffused reduction in structural integrity of the gastrointestinal tract (e.g. peptic ulcer, acute diverticulitis)
* severe hepatic insufficiency (Child-Pugh Class C)
* renal impairment (glomerular filtration rate < 90 ml/min) with or without renal replacement therapy
* severe diarrhea despite high opioid dosing
* participation in another study with an investigational drug within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of methylnaltrexone (Cmax, tmax, area under the curve, total clearance, halflife, accumulation ratio, renal clearance) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Natascia Corti, MD, Principal Investigator — University Hospital Zurich, Pharmacology and Toxicology
Locations (1):
- Neurointensive Care Unit, Zurich, Switzerland